CLINICAL TRIAL: NCT02281136
Title: A Pharmacokinetic Study of Levulan Kerastick (Aminolevulinic Acid HCl) for Topical Solution, 20% Under Maximal Use Conditions
Brief Title: Maximal Use Systemic Exposure (MUSE) Study of Levulan Kerastick
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CP0110
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Keratosis, Actinic
Keywords: Actinic keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALA (Experimental): 20% aminolevulinic acid applied via Kerastick to individual AK lesions on the upper extremities and covered with occlusive dressing for 3 hours prior to BLU-U treatment
  Interventions: Drug: Aminolevulinic Acid (ALA); Device: BLU-U

INTERVENTIONS:
Drug: Aminolevulinic Acid (ALA) — 20% ALA applied to upper extremities for 3 hours prior to 10 J/cm2 blue light
  Other Names: Levulan Kerastick
Device: BLU-U — 10 J/cm2 of 417 nm blue light delivered at 10 mW/cm2
  Other Names: Blue Light Photodynamic Therapy (PDT)

SUMMARY:
The purpose of this study is to evaluate the potential for systemic exposure of aminolevulinic acid (ALA) when applied topically under occlusion, in a maximal use setting in patients with multiple actinic keratoses (AK) involving the upper extremities.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 Grade 1/2 AKs on one upper extremity AND
* At least 12 Grade 1/2 AKs on the OTHER upper extremity

Exclusion Criteria:

* Pregnancy
* history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins or photodermatosis
* lesions suspicious for skin cancer (skin cancer not ruled out by biopsy) or untreated skin cancers within the Treatment Area
* Body Mass Index (BMI) > 32.0 kg/m2
* skin pathology or condition which could interfere with the evaluation of the test product or requires the use of interfering topical or systemic therapy
* significant blood loss within 60 days or donated blood/plasma within 72 hours prior to Visit 2 (Baseline)
* tested positive at screening for human immunodeficiency virus (HIV) or was known to be seropositive for HIV
* a history of lead poisoning or a history of a significant exposure to lead or a screening lead level above 6μg/dl
* tested positive at screening for hepatitis B surface antigen, hepatitis C antibody or had a history of a positive result
* positive drug screen at Screening
* Screening safety labs are clinically significant in the opinion of the investigator
* major surgery within 30 days prior to Visit 2 (Baseline) or plans to have surgery during the study
* Subject is immunosuppressed
* currently enrolled in an investigational drug or device study
* has received an investigational drug or been treated with an investigational device within 30 days prior to Visit 2 (Baseline)
* known sensitivity to one or more of the vehicle components (ethyl alcohol, isopropyl alcohol, laureth 4, polyethylene glycol)
* use of the following topical preparations on the extremities to be treated:

  * Keratolytics including urea (greater than 5%), alpha hydroxyacids [e.g.glycolic acid, lactic acid, etc. greater than 5%], salicylic acid (greater than 2%) within 2 days of initiation of treatment
  * Cryotherapy within 2 weeks of initiation of treatment
  * Retinoids, including tazarotene, adapalene, tretinoin, retinol, within 4 weeks of initiation of treatment
  * Microdermabrasion, laser ablative treatments, ALA-PDT, chemical peels, 5-FU, diclofenac, imiquimod or other topical treatments for AK within 8 weeks of initiation of treatment
* use of systemic retinoid therapy within 6 months of initiation of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Marcus, MD, PhD, Study Director — DUSA Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Therapeutics Clinical Research, San Diego, California
  - Shideler Clinical Research Center, Carmel, Indiana
  - DermResearch, Inc., Austin, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Levulan Kerastick: 20% aminolevulinic acid applied via Kerastick to individual AK lesions on the upper extremities and covered with occlusive dressing for 3 hours prior to BLU-U treatment
  Aminolevulinic Acid (ALA): 20% ALA applied to upper extremities for 3 hours prior to 10 J/cm2 blue light
  BLU-U: 10 J/cm2 of 417 nm blue light delivered at 10 mW/cm2
Period: Overall Study
Arm/Group | Levulan Kerastick
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (8.8)
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Maximum Baseline Corrected Plasma Concentration (Cmax) for ALA
Description: Maximum baseline corrected plasma concentration (Cmax) for ALA over the 24 hour sampling time period. Blood samples wiere taken before ALA application and at 15 and 30 minutes, 1, 2, 4, 8, 12, 16 and 24 hours following study medication application.
Time Frame: 1 day
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
ng/mL | 79.85 (221.7)

2. Primary Outcome: Time at Which Cmax is Attained (Tmax) for ALA
Description: Time of the maximum baseline corrected plasma concentration for ALA measured at at 15 and 30 minutes, 1, 2, 4, 8, 12, 16 and 24 hours following study medication application.If a maximum value occurred at more than one timepoint Tmax is defined as the first timepoint with this value.
Time Frame: 1 day
Measure: Median (Full Range); unit: hours
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
hours | 2 [0.25 to 4.05]

3. Primary Outcome: AUCt
Description: AUCt is the area under the baseline corrected plasma concentration-time profile up to the last quantifiable/non-negative plasma concentration
Time Frame: 0, 15, 30 minutes, and 1, 2, 4, 8, 12, 16, 24 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
ng*hr/mL | 282.1 (163)

4. Primary Outcome: The Terminal Exponential Half-life (T1/2,z)
Description: The terminal slope will be calculated by linear least squares regression of the log plasma concentration-time data. The terminal exponential half-life (T1/2,z) will be calculated as 0.693 divided by the absolute value of slope.
Time Frame: 1 day
Population: T1/2,z could not be determined in 4 subjects
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 25
hours | 4.602 (78.83)

5. Secondary Outcome: Hyperpigmentation
Description: HYPERPIGMENTATION SCALE Grade 0 = No hyperpigmentation Grade 1 = Light hyperpigmentation involving small areas Grade 2 = Moderate hyperpigmentation involving small areas; light hyperpigmentation involving moderate areas Grade 3 = Moderate hyperpigmentation involving moderate sized areas; light hyperpigmentation involving large areas; small areas of marked hyperpigmentation Grade 4 = Marked hyperpigmentation involving moderate or large sized areas
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 7
  Grade 1 | 14
  Grade 2 | 5
  Grade 3 | 3
  Grade 4 | 0

6. Secondary Outcome: Hyperpigmentation
Description: as for outcome 5
Time Frame: 24 hours after PDT
Population: One subject did not have assessment performed
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 28
participants
  Grade 0 | 6
  Grade 1 | 14
  Grade 2 | 4
  Grade 3 | 4
  Grade 4 | 0

7. Secondary Outcome: Hyperpigmentation
Description: as for outcome 5
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 6
  Grade 1 | 14
  Grade 2 | 6
  Grade 3 | 3
  Grade 4 | 0

8. Secondary Outcome: Hypopigmentation
Description: HYPOPIGMENTATION SCALE Grade 0 = No hypopigmentation Grade 1 = Light hypopigmentation involving small areas Grade 2 = Moderate hypopigmentation involving small areas; light hypopigmentation involving moderate areas Grade 3 = Moderate hypopigmentation involving moderate sized areas; light hypopigmentation involving large areas; small areas of marked hypopigmentation Grade 4 = Marked hypopigmentation involving moderate or large sized areas
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 10
  Grade 1 | 16
  Grade 2 | 3
  Grade 3 | 0
  Grade 4 | 0

9. Secondary Outcome: Hypopigmentation
Description: as for outcome 8
Time Frame: 24 hours post PDT#1
Population: One subject did not have assessment performed
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 28
participants
  Grade 0 | 9
  Grade 1 | 18
  Grade 2 | 0
  Grade 3 | 1
  Grade 4 | 0

10. Secondary Outcome: Hypopigmentation
Description: as for outcome 8
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 8
  Grade 1 | 21
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

11. Secondary Outcome: Erythema
Description: Erythema Scale - Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 23
  Grade 1 | 6
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

12. Secondary Outcome: Erythema
Description: as for outcome 11
Time Frame: 5 Minutes after PDT
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 0
  Grade 1 | 0
  Grade 2 | 7
  Grade 3 | 19
  Grade 4 | 3

13. Secondary Outcome: Erythema
Description: as for outcome 11
Time Frame: 24 hours after PDT #1
Population: One subject did not have assessment performed
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 28
participants
  Grade 0 | 4
  Grade 1 | 0
  Grade 2 | 9
  Grade 3 | 13
  Grade 4 | 2

14. Secondary Outcome: Erythema
Description: as for outcome 11
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 12
  Grade 1 | 7
  Grade 2 | 10
  Grade 3 | 0
  Grade 4 | 0

15. Secondary Outcome: Edema
Description: EDEMA SCALE Grade 0 = None Grade 1 = Minimal - scant, rare edema Grade 2 = Mild - easily seen edema, minimally palpable, involving up to 1/3 of the treatment area Grade 3 = Moderate - easily seen edema and typically palpable, involving between 1/3 to 2/3 of the treatment area Grade 4 = Severe - easily seen edema, indurated in some areas, involving over 2/3 of the treatment area
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 29
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

16. Secondary Outcome: Edema
Description: as for outcome 15
Time Frame: 5 Minutes after PDT
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 22
  Grade 1 | 3
  Grade 2 | 2
  Grade 3 | 2
  Grade 4 | 0

17. Secondary Outcome: Edema
Description: as for outcome 15
Time Frame: 24 hours after PDT #1
Population: One subject did not have assessment performed
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 28
participants
  Grade 0 | 22
  Grade 1 | 4
  Grade 2 | 2
  Grade 3 | 0
  Grade 4 | 0

18. Secondary Outcome: Edema
Description: as for outcome 15
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 29
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

19. Secondary Outcome: Stinging/Burning
Description: STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 29
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 0

20. Secondary Outcome: Stinging/Burning
Description: as for outcome 19
Time Frame: During PDT
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 0
  Grade 1 | 0
  Grade 2 | 19
  Grade 3 | 10

21. Secondary Outcome: Stinging/Burning
Description: as for outcome 19
Time Frame: 5 Minutes after PDT
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 0
  Grade 1 | 21
  Grade 2 | 7
  Grade 3 | 1

22. Secondary Outcome: Stinging/Burning
Description: as for outcome 19
Time Frame: 24 hours after PDT #1
Population: One subject did not have assessment performed
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 28
participants
  Grade 0 | 18
  Grade 1 | 9
  Grade 2 | 1
  Grade 3 | 0

23. Secondary Outcome: Stinging/Burning
Description: as for outcome 19
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 29
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 0

24. Secondary Outcome: Scaling and Dryness
Description: SCALING AND DRYNESS SCALE Grade 0 = None Grade 1 = Minimal - barely perceptible desquamation Grade 2 = Mild - limited areas of fine desquamation in up to 1/3 of the treatment area Grade 3 = Moderate - fine desquamation involving 1/3 to 2/3 of the treatment area or limited areas of coarser scaling Grade 4 = Severe - coarser scaling involving more than 2/3 of the treatment area or limited areas of very coarse scaling
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 25
  Grade 1 | 1
  Grade 2 | 3
  Grade 3 | 0
  Grade 4 | 0

25. Secondary Outcome: Scaling and Dryness
Description: as for outcome 24
Time Frame: 24 hours after PDT #1
Population: One subject did not have assessment performed
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 28
participants
  Grade 0 | 20
  Grade 1 | 7
  Grade 2 | 1
  Grade 3 | 0
  Grade 4 | 0

26. Secondary Outcome: Scaling and Dryness
Description: as for outcome 24
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 19
  Grade 1 | 9
  Grade 2 | 1
  Grade 3 | 0
  Grade 4 | 0

27. Secondary Outcome: OOZING/VESICULATION/CRUSTING
Description: OOZING/VESICULATION/CRUSTING Grade 0 = None Grade 1 = Minimal - a single area of oozing, vesiculation or crusting 3 mm diameter or less in size Grade 2 = Mild - two to four areas of oozing, vesiculation or crusting 3 mm diameter or less in size OR a single area larger than 3 mm diameter in size Grade 3 = Moderate - more than a single area of oozing, vesiculation or crusting larger than 3 mm diameter in size or more than four areas of 3 mm diameter or less in size Grade 4 = Severe - any degree of oozing, vesiculation or crusting greater than (3) above
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 29
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

28. Secondary Outcome: OOZING/VESICULATION/CRUSTING
Description: as for outcome 27
Time Frame: 24 hours after PDT #1
Population: One subject did not have assessment performed
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 28
participants
  Grade 0 | 27
  Grade 1 | 1
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

29. Secondary Outcome: OOZING/VESICULATION/CRUSTING
Description: as for outcome 27
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | Levulan Kerastick
Number analyzed (Participants) | 29
participants
  Grade 0 | 28
  Grade 1 | 1
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Levulan Kerastick
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 1/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levulan Kerastick (N=29)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication of results will be made by the Sponsor. If publication is not submitted within 12 months after the date of study final report, the PI may publish the results from the site individually, subject to compliance with the other terms of the clinical trial agreement, including a requirement that the PI provide a draft of the publication for the sponsor's review 30 days before submission for publication so that sponsor can review the publication for confidential information